CLINICAL TRIAL: NCT07011862
Title: COBRA: Cancer, Older Adults, Balance and Resistance Activities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-090
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Primary Cancer; Metastatic Cancer; Cancer
Keywords: Primary Cancer; Metastatic Cancer; Cancer; 25-090; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older Adult Patients/OAP (Experimental): Older Adult Patients with Cancer are within 1 year of completion of primary therapy for cancer OR have a diagnosis of metastatic cancer;
  Interventions: Behavioral: Cancer, Older adults, Balance and Resistance Activities

INTERVENTIONS:
Behavioral: Cancer, Older adults, Balance and Resistance Activities — The COBRA intervention is delivered as a web-based application through an iPad configured to allow access only to the study application and Zoom videoconferencing icons during the trial.
  Other Names: COBRA

SUMMARY:
The purpose of this study is to find out whether an 8-week digital health promotion program called COBRA is a safe and practical (feasible) option for older adults with cancer/OAC.

ELIGIBILITY:
Inclusion Criteria:

Older Adult Patients with Cancer

- Are within 1 year of completion of primary therapy for cancer OR have a diagnosis of metastatic cancer;

1. For the purpose of this study, primary therapy is defined as treatment of curative intent, first-line or later, from which the individual is advancing to active surveillance or follow-up with or without maintenance therapy.
2. Individuals with metastatic cancer may be included provided they have stable disease or better per most recent restaging exam at time of enrollment.

i. Patients with stable metastatic bony disease at most recent restaging exam and a score of 0-2 on the Functional Pain Scale (FPS69; Appendix 18) are eligible. The PI will consult with the Rehab Med co-PI for FPS scores of 3 or greater, by patient request or PI discretion.

ii. Patients with symptomatic visceral metastases will be evaluated on a case-by-case basis at time of enrollment.

* Are aged 65 years and older, with no upper age limit;
* ECOG PS 0-3 or Karnofsky PS greater than or equal to 40;
* Can read and speak English;
* Self-report access to internet connection sufficient to support videoconferencing.

Clinicians

* Licensed clinician (MD, RN, APP) with an interest in the care of older adults with cancer.

Exclusion Criteria:

Older Adult Patients with Cancer

* Have any cognitive impairment, neurologic, musculoskeletal, or other comorbid condition (as assessed by their provider) that would prevent the individual from engaging with the digital health coaching program or complete study assessments or engage in progressive intensity levels of physical activity
* Have a neurologic, musculoskeletal, or other comorbid condition that would impede their ability to safely engage in progressive intensity levels of physical activity (as assessed by their provider). Patients with metastatic disease and suspected interim progression since last restaging exam will be referred back to their primary oncology care team for evaluation prior to enrollment.
* Have activity restrictions post-surgery at the time of enrollment

Clinicians No expected exclusions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of retention and adherence to the COBRA/Cancer, Older Adults, Balance and Resistance Activities intervention | 8 weeks
  Rate of retention and adherence to the 8-week intervention to define intervention feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Fessele, PhD, RN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org